CLINICAL TRIAL: NCT01998282
Title: Assessing the Impact of Water Filters and Improved Cook Stoves on Drinking Water and Quality and Indoor Air Pollution: A Matched Cohort Study in Rwanda
Brief Title: Evaluation of a Project to Distribute Water Filters and Cook Stoves in Western Rwanda--Phase 1B
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Ministry of Health, Rwanda (Other Government); DelAgua (Other); Portland State University (Other); University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Thomas Clasen, Reader in Water, Sanitation and Health, London School of Hygiene and Tropical Medicine
Other Study IDs: 6457
Record Dates: First submitted 2013-11-08; First posted 2013-11-28 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Focus of Study is to Assess Filter and Stove Use and Efficacy in Reducing Exposure to Waterborne and Airborne Pathogens
Keywords: Focus of study is to assess filter/stove use and efficacy in reducing exposure to waterborne and airborne pathogens.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Household water filter and improved cook stove: Vestergaard-Frandsen LifeStraw Family 2.0 filter and Ecozoom stove
- Control: Traditional water management practices and cooking stoves

SUMMARY:
DelAgua Health and Development, Manna Energy and the Rwanda Ministry of Health are collaborating on a project financed by carbon credits that will distribute household-based water filters and high-efficiency cook stoves to approximately 600,000 households in Rwanda. Prior to the full roll out of the campaign, the implementers are conducting research in connection with a distribution among 2000 households in western Rwanda. The objective of this matched cohort study (Phase 1B)are to investigate whether the filters and stoves delivered in October 2012 are still performing and in use, to determine whether they are associated with reductions in exposure to pathogens from drinking water and stoves, and to assembly information on health and other conditions necessary for the design of a large scale health impact evaluation.

ELIGIBILITY:
Households will be eligible to participate in the study if they reside in selected villages and are willing to participate after receiving complete details regarding the study. Intervention households must have a functioning stove and water filter in order to participate, though they do not need to be in regular use. We will enroll all households with a child under 5 years of age if they are in Ubudehe groups 1 or 2.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lower income (ubudehe groups 1 and 2) householders from 18 villages (9 intervention and matched controls) in 11 designated Districts in Rwanda: Rutsiro, Karongi, Ngororero, Nyamasheke, Nyabihu Districts of Western Province (excluding part of the district to the north of the Ruhengeri road); Rubuvu District (excluding part of the district to the north of the Ruhengeri road); Nyaruguru, Nyamagabe, Muhanga, and Ruhango Districts in Southern Province; Gakenke District in Northern Province.
Sampling Method: Probability Sample
Enrollment: 1035 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Personal exposure to PM2.5 and CO (mg/m3) | 10 months
  PM2.5 and CO concentrations will be measure in mg/m3 and reported as the mean concentration over 48 hours.

SECONDARY OUTCOMES:
Thermotolerant coliforms (TTC) in colony forming units (CFU) per 100ml of sample water | 10 months
  TTC will be measured as the total number of colony forming units (CFU) of TTC in the water sample and will be reported as number of CFU per 100ml of sample water.

OTHER OUTCOMES:
Blood pressure | 10 months
Blood pressure covariates | 10 months
Use of filter and stove | 10 months
Exposure to PM2.5 and CO in primary cooking areas (mg/m3) | 10 months
  PM2.5 and CO concentrations during the 48 hour sampling period

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Clasen, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- DelAgua Health Rwanda, Kigali, PO Box 1594, Rwanda